CLINICAL TRIAL: NCT06636188
Title: Novel Artificial Intelligence Patient Navigator Chatbot to Reduce Physical and Psychological Distress of Patients With Head and Neck Cancer Undergoing Radiotherapy: A Randomized Controlled Trial
Brief Title: A Chatbot to Reduce Physical and Psychological Distress of Patients With Head and Neck Cancer Undergoing Radiotherapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Tongyao WANG, Research Assitant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KC/KE-23-0116/ER-4
Record Dates: First submitted 2024-10-03; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer
Keywords: chatbot; digital health; oncology care
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-As-Usual Arm (No Intervention): Participants in the Treatment-As-Usual group will receive routine onsite nursing care in which the nurse discusses general knowledge of self-care behaviors regarding the management of radiotherapy-related side effects.
- Digi-Coach Chatbot Arm (Experimental): Participants in Digi-Coach Chatbot Arm will have access to the Digi-Coach chatbot in addition to usual care. The research nurse will provide training on how to use the chatbot.
  Interventions: Other: Digi-Coach Chatbot

INTERVENTIONS:
Other: Digi-Coach Chatbot — Participants will have access to the Digi-Coach chatbot in addition to usual care. The research nurse will provide training on how to navigate the chatbot and ask participants to query all their cancer related concerns in the chatbot.
  Arms: Digi-Coach Chatbot Arm

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of the Digi-Coach chatbot for reducing physical and psychological distress in people undergoing radiotherapy for head and neck cancer.

The main question it aims to answer is: How effective is the Digi-Coach chatbot in reducing physical and psychological distress?

Researchers will compare Digi-Coach chatbot to usual nursing care to see if Digi-Coach chatbot is effective for reducing physical and psychological distress in people undergoing radiotherapy for head and neck cancer.

Participants will have access to the Digi-Coach chatbot during radiotherapy in addition to usual care. The research nurse will provide training on how to navigate the chatbot and ask participants to query all their cancer-related concerns in the chatbot.

DETAILED DESCRIPTION:
The goal of this clinical trial is to assess the effectiveness of the Digi-Coach chatbot for reducing physical and psychological distress in people undergoing radiotherapy for head and neck cancer.

The main question it aims to answer is: How effective is the Digi-Coach chatbot in reducing physical and psychological distress? Researchers will compare Digi-Coach chatbot to usual nursing care to see if Digi-Coach chatbot is effective for reducing physical and psychological distress in people undergoing radiotherapy for head and neck cancer.

A single-blinded parallel randomized controlled trial (RCT allocation ratio = 1:1) will be conducted, with baseline data collection at week 1 (T0) and three follow-up timepoints at week 8 (T1), week 12 (T2) following radiotherapy commencement.

Participants in the Treatment-As-Usual group will receive routine onsite nursing care in which the nurse discussed general knowledge of self-care behaviors regarding the management of radiotherapy-related side effects.

Participants in the intervention group will have access to the Digi-Coach chatbot in addition to usual care. The research nurse will provide training on how to navigate the chatbot and ask participants to query all their cancer-related concerns in the chatbot.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 and above
* are able to read and speak Cantonese or Mandarin fluently
* have a new, primary diagnosis of head and neck/laryngeal cancer
* are waiting to receive a full course of curative-intent, external beam radiotherapy with or without chemotherapy
* have a Karnofsky performance score ≥70
* have distress scored 3 or above on the NCCN distress thermometer

Exclusion Criteria:

* insufficient command of Chinese
* have any other factors precluding the ability to give informed consent or comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
National Comprehensive Cancer Network Distress Thermometer | 1 week, 8 weeks, and 12 weeks
  A 2-item measurement that has participants first rate their distress levels on a scale of 0 (no distress) to 10 (extreme distress) and then self-report their concerns by choosing from a given list of physical, emotional, social, practical, spiritual, or other concerns.

SECONDARY OUTCOMES:
Memorial Symptom Assessment Scale | 1 week, 8 weeks, and 12 weeks
  32-item comprehensive tool for assessing cancer-related symptom burden with three analysis domains of symptom severity (1 = slight, 4 = very severe), prevalence (1 = rarely, 4 = almost constantly), and distress (0 = not at all, 4 = very much).
Functional Assessment of Cancer Therapy-Head and Neck | 1 week, 8 weeks, and 12 weeks
  27 items on the general well-being domain (physical, social/family, emotional, and functional) and 11 items specific to head and neck cancer on a 5-point Likert scale. The total score ranges from 0 to 148; the higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tongyao Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The de-identified individual participant data will not be shared, as the participants did not consent to their data being shared with others at the time of collection.